CLINICAL TRIAL: NCT03800719
Title: Personalized Support Using Instant Messaging Applications to Increase Smoking Cessation in Smokers Proactively Recruited From Smoking Hotspots in Hong Kong: a Pragmatic Randomized Controlled Trial
Brief Title: Personalized Support Using Instant Messaging Applications to Increase Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Personalized IM+referral
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; active referral; IM
MeSH Terms: conditions — Smoking Cessation | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): AWARD advice, health warning leaflet, active referral to smoking cessation (SC) services, regular messages through Instant Messaging (IM), psychosocial support and referral to SC services through IM
  Interventions: Behavioral: AWARD advice; Behavioral: Health warning leaflet; Behavioral: Active referral to smoking cessation (SC) services; Behavioral: Regular messages through Instant Messaging (IM); Behavioral: Psychosocial support and referral to SC services through IM
- Control Group (Active Comparator): AWARD advice, health warning leaflet, active referral to smoking cessation (SC) services, SMS message on general health
  Interventions: Behavioral: AWARD advice; Behavioral: Health warning leaflet; Behavioral: Active referral to smoking cessation (SC) services; Behavioral: Message on general health delivered by short message service (SMS)

INTERVENTIONS:
Behavioral: AWARD advice — At baseline, brief smoking cessation advice following AWARD model will be delivered to subjects within about 2 to 5 minutes:
  * Ask about smoking history and habit
  * Warn about the risks of smoking using a leaflet
  * Advise to quit smoking as soon as possible and use nicotine replacement therapy (NRT) or SC services
  * Refer subjects to free smoking cessation services in Hong Kong if they agree
  * Do it again: smokers who have tried to quit but relapsed will be encouraged to quit again and those who have reduced smoking will be advised to further reduce or quit smoking
Behavioral: Health warning leaflet — At baseline, an A5-sized leaflet will be given to subjects, which includes information about risks of smoking, pictures of smoking-related diseases, and smoking cessation services provided in Hong Kong.
Behavioral: Active referral to smoking cessation (SC) services — At baseline, subjects will be encouraged to seek smoking cessation services in Hong Kong. If subjects agree, their contact information will be sent to the preferred service providers for a quick appointment and follow-up.
Behavioral: Regular messages through Instant Messaging (IM) — A total of pre-set 26 messages will be sent to subjects through WhatsApp 12 weeks after baseline to remind the quit date and to encourage abstinence. Messages are tailored based on subjects' sociodemographic characteristics and smoking habit following Social Cognitive Theory and Transtheoretical Model. Messages will be sent with the schedule of once daily for 1 week (the week across the quit date), 3 times a week for 4 weeks (2 weeks each before and after the week with quit date) and once a week for remaining 7 weeks. The schedule will be adjusted according to the quit date and also smokers' requests. The format of regular messages will mainly be text-based but also include pictures, animations and videos.
  Arms: Intervention Group
Behavioral: Psychosocial support and referral to SC services through IM — Personalized interactive text or voice conversation will be provided by trained smoking cessation advisors through WhatsApp for 3 months after baseline. Advisors will periodically proactively send messages to subjects to initiate the conversation (e.g. asking recent progress of smoking cessation) and deliver evidence-based advice. Advisors will also actively refer subjects, if they have expressed the need, to smoking cessation services providers. A standard operation algorithm for advisors used in the pilot feasibility trial will be modified for the use.
  Arms: Intervention Group
Behavioral: Message on general health delivered by short message service (SMS) — After baseline, regular messages using SMS will be sent to subjects with similar frequency to Intervention group. The messages include information on general health and reminders on follow-up surveys and biochemical validation for quitting.
  Arms: Control Group

SUMMARY:
This study aims to assess the effect of personalized support using instant messaging application on smoking cessation in smokers proactively recruited from smoking hotspots in Hong Kong.

DETAILED DESCRIPTION:
Detailed Description: With the advancement of information communication technologies (ICTs), instant messaging applications (IM Apps, e.g. WhatsApp and WeChat) can be used for providing synchronous, personalized, interactive interventions for health promotion. This study proposes to apply IM Apps for enhancing our tested brief smoking cessation (SC) intervention model from AWARD to e-AWARD (AWARD: Ask, Warn, Advise, Refer, Do-it-again,) without medications to increase SC in smokers proactively recruited in smoking hotspots in Hong Kong. Such smokers are the majority and have low quit rate. IM Apps allows trained SC advisors to proactively deliver personalized SC advices, response to smokers' needs promptly, and provide psychosocial support. No similar trials are found in PubMed, Cochrane Library and trial registries (ClinicalTrials.gov & ISRCTN) (except the pilot trial of this study). The aims of this study are as follows:

1. To assess the main effect of the personalized support using instant messaging applications (Intervention) vs. Control group on biochemical validated smoking abstinence at 6-month and 12-month.
2. To assess the effects on self-reported past 7-day abstinence, 24-week continuous abstinence, smoking reduction, self-efficacy of quitting, intention to quit, quit attempts and SC medications and services use at 6-month and 12-month.
3. To identify the mediators, which can inform mechanisms of the intervention on SC.
4. To evaluate the cost-effectiveness of the above interventions.
5. To understand the effects subjects' experience of IM support on SC using a qualitative study approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult smokers aged 18+ who smoke cigarette(s) daily.
* Exhaled carbon monoxide (CO) level of 4ppm or above.
* Having smartphones with IM Apps (WhatsApp) and have experience in using.
* Hong Kong residents able to read and communicate in Chinese (Cantonese or Putonghua).

Exclusion Criteria:

* Smokers who have psychiatric/psychological diseases or are on regular psychotropic medications.
* Smokers who are using SC medication, NRT, other SC services or projects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 696 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically-validated abstinence at 6-month | 6-month after baseline
  Defined as exhaled carbon monoxide <4ppm
Biochemically-validated abstinence at 12-month | 12-month after baseline
  Defined as exhaled carbon monoxide <4ppm

SECONDARY OUTCOMES:
Self-reported past 7-day abstinence | 6-month and 12-month after baseline
  Self-reported no cigarette smoking (even a single puff) in the past 7 days
Self-reported 24-week continuous abstinence | 6-month and 12-month after baseline
  Self-reported no cigarette smoking (even a single puff) in the past 24 weeks
Smoking reduction | 6-month and 12-month after baseline
  Self-reported reduction in the number of cigarettes smoked daily by at least 50% of the baseline amount
Perceived importance, confidence and difficulties of quitting | 6-month and 12-month after baseline
  Perceived importance, confidence and difficulties of quitting measured on a scale of 0-10 and a higher score indicates a stronger perception
Intention to quit | 6-month and 12-month after baseline
  Any intention to quit smoking (yes/no) from baseline
Quit attempts | 6-month and 12-month after baseline
  Number of quit attempts from baseline
Smoking cessation medication use | 6-month and 12-month after baseline
  Any use of nicotine replacement therapy from baseline
Smocking cessation services use | 6-month and 12-month after baseline
  Any use of counselling, hotline, SC clinics and other SC services from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Lam TH, Cheung YT, Leung DY, Abdullah AS, Chan SS. Effectiveness of smoking reduction intervention for hardcore smokers. Tob Induc Dis. 2015 Apr 2;13(1):9. doi: 10.1186/s12971-015-0034-y. eCollection 2015. PMID 25859176
- [Background] Census and Statistics Department. Thematic Household Survey, Report No.59: Pattern of Smoking Hong Kong SAR: Hong Kong SAR Government. 2016. Available from: http://www.statistics.gov.hk/pub/B11302592016XXXXB0100.pdf.
- [Background] Aveyard P, Begh R, Parsons A, West R. Brief opportunistic smoking cessation interventions: a systematic review and meta-analysis to compare advice to quit and offer of assistance. Addiction. 2012 Jun;107(6):1066-73. doi: 10.1111/j.1360-0443.2011.03770.x. Epub 2012 Feb 28. PMID 22175545
- [Background] Chan SS, Wong DC, Cheung YT, Leung DY, Lau L, Lai V, Lam TH. A block randomized controlled trial of a brief smoking cessation counselling and advice through short message service on participants who joined the Quit to Win Contest in Hong Kong. Health Educ Res. 2015 Aug;30(4):609-21. doi: 10.1093/her/cyv023. Epub 2015 Jun 25. PMID 26116584
- [Background] Chan SSC, Cheung YTD, Wan Z, Wang MP, Lam TH. Proactive and Brief Smoking Cessation Intervention for Smokers at Outdoor Smoking "Hotspots" in Hong Kong. J Cancer Educ. 2018 Apr;33(2):365-370. doi: 10.1007/s13187-016-1085-3. PMID 27474113
- [Background] Wang MP, Li WH, Cheung YT, Lam OB, Wu Y, Kwong AC, Lai VW, Chan SS, Lam TH. Brief Advice on Smoking Reduction Versus Abrupt Quitting for Smoking Cessation in Chinese Smokers: A Cluster Randomized Controlled Trial. Nicotine Tob Res. 2017 Dec 13;20(1):67-72. doi: 10.1093/ntr/ntx026. PMID 28182243
- [Background] Cheung YT, Wang MP, Li HC, Kwong A, Lai V, Chan SS, Lam TH. Effectiveness of a small cash incentive on abstinence and use of cessation aids for adult smokers: A randomized controlled trial. Addict Behav. 2017 Mar;66:17-25. doi: 10.1016/j.addbeh.2016.11.006. Epub 2016 Nov 10. PMID 27863323
- [Background] Chan SSC, Cheung YTD, Wong YMB, Kwong A, Lai V, Lam TH. A Brief Smoking Cessation Advice by Youth Counselors for the Smokers in the Hong Kong Quit to Win Contest 2010: a Cluster Randomized Controlled Trial. Prev Sci. 2018 Feb;19(2):209-219. doi: 10.1007/s11121-017-0823-z. PMID 28755244
- [Background] Cheung YTD, Lam TH, Li WHC, Wang MP, Chan SSC. Feasibility, Efficacy, and Cost Analysis of Promoting Smoking Cessation at Outdoor Smoking "Hotspots": A Pre-Post Study. Nicotine Tob Res. 2018 Nov 15;20(12):1519-1524. doi: 10.1093/ntr/ntx147. PMID 28655173
- [Background] Wang MP, Suen YN, Li WH, Lam CO, Wu SY, Kwong AC, Lai VW, Chan SS, Lam TH. Intervention With Brief Cessation Advice Plus Active Referral for Proactively Recruited Community Smokers: A Pragmatic Cluster Randomized Clinical Trial. JAMA Intern Med. 2017 Dec 1;177(12):1790-1797. doi: 10.1001/jamainternmed.2017.5793. PMID 29059277
- [Background] Wright J. Very brief advice can be effective in encouraging smokers to quit 2013 Available from: http://www.guidelinesinpractice.co.uk/jan_13_wright_smoking_jan13#.Vf927RGqqko.
- [Background] Free C, Knight R, Robertson S, Whittaker R, Edwards P, Zhou W, Rodgers A, Cairns J, Kenward MG, Roberts I. Smoking cessation support delivered via mobile phone text messaging (txt2stop): a single-blind, randomised trial. Lancet. 2011 Jul 2;378(9785):49-55. doi: 10.1016/S0140-6736(11)60701-0. PMID 21722952
- [Background] Abroms LC, Boal AL, Simmens SJ, Mendel JA, Windsor RA. A randomized trial of Text2Quit: a text messaging program for smoking cessation. Am J Prev Med. 2014 Sep;47(3):242-50. doi: 10.1016/j.amepre.2014.04.010. Epub 2014 Jun 6. PMID 24913220
- [Background] Naughton F, Cooper S, Foster K, Emery J, Leonardi-Bee J, Sutton S, Jones M, Ussher M, Whitemore R, Leighton M, Montgomery A, Parrott S, Coleman T. Large multi-centre pilot randomized controlled trial testing a low-cost, tailored, self-help smoking cessation text message intervention for pregnant smokers (MiQuit). Addiction. 2017 Jul;112(7):1238-1249. doi: 10.1111/add.13802. Epub 2017 May 2. PMID 28239919
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Apr 10;4(4):CD006611. doi: 10.1002/14651858.CD006611.pub4. PMID 27060875
- [Background] Scott-Sheldon LA, Lantini R, Jennings EG, Thind H, Rosen RK, Salmoirago-Blotcher E, Bock BC. Text Messaging-Based Interventions for Smoking Cessation: A Systematic Review and Meta-Analysis. JMIR Mhealth Uhealth. 2016 May 20;4(2):e49. doi: 10.2196/mhealth.5436. PMID 27207211
- [Background] Hoeppner BB, Hoeppner SS, Abroms LC. How do text-messaging smoking cessation interventions confer benefit? A multiple mediation analysis of Text2Quit. Addiction. 2017 Apr;112(4):673-682. doi: 10.1111/add.13685. Epub 2016 Dec 12. PMID 27943511
- [Background] Douglas N, Free C. 'Someone batting in my corner': experiences of smoking-cessation support via text message. Br J Gen Pract. 2013 Nov;63(616):e768-76. doi: 10.3399/bjgp13X674459. PMID 24267860
- [Background] Hoermann S, McCabe KL, Milne DN, Calvo RA. Application of Synchronous Text-Based Dialogue Systems in Mental Health Interventions: Systematic Review. J Med Internet Res. 2017 Jul 21;19(8):e267. doi: 10.2196/jmir.7023. PMID 28784594
- [Background] Hamine S, Gerth-Guyette E, Faulx D, Green BB, Ginsburg AS. Impact of mHealth chronic disease management on treatment adherence and patient outcomes: a systematic review. J Med Internet Res. 2015 Feb 24;17(2):e52. doi: 10.2196/jmir.3951. PMID 25803266
- [Background] Wang MP, Li WH, Jiang N, Chu LY, Kwong A, Lai V, Lam TH. E-Cigarette Awareness, Perceptions and Use among Community-Recruited Smokers in Hong Kong. PLoS One. 2015 Oct 26;10(10):e0141683. doi: 10.1371/journal.pone.0141683. eCollection 2015. PMID 26502284
- [Background] Lindson-Hawley N, Thompson TP, Begh R. Motivational interviewing for smoking cessation. Cochrane Database Syst Rev. 2015 Mar 2;(3):CD006936. doi: 10.1002/14651858.CD006936.pub3. PMID 25726920
- [Background] Stead LF, Hartmann-Boyce J, Perera R, Lancaster T. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2013 Aug 12;(8):CD002850. doi: 10.1002/14651858.CD002850.pub3. PMID 23934971
- [Background] Thematic household survey Report No.62: Information technology usage and penetration. Hong Kong SAR Government. 2016. Available from: http://www.digital21.gov.hk/eng/statistics/download/informationsociety2013.pdf. 25. Bandura A.
- [Background] Social Foundation of Thought and Action: A Social Cognitive Theory. Englewood Cliffs, NJ: Prentice-Hall; 1986.
- [Background] Department of Health. Smoking Cessation Information Kit. Hong Kong SAR: 2015. Avialabe from: https://www.tco.gov.hk/english/quitting/files/kit09_eng.pdf
- [Background] Cheung YT, Chan CH, Lai CK, Chan WF, Wang MP, Li HC, Chan SS, Lam TH. Using WhatsApp and Facebook Online Social Groups for Smoking Relapse Prevention for Recent Quitters: A Pilot Pragmatic Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Oct 22;17(10):e238. doi: 10.2196/jmir.4829. PMID 26494159
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Chan SS, Leung DY, Wong DC, Lau CP, Wong VT, Lam TH. A randomized controlled trial of stage-matched intervention for smoking cessation in cardiac out-patients. Addiction. 2012 Apr;107(4):829-37. doi: 10.1111/j.1360-0443.2011.03733.x. Epub 2012 Jan 23. PMID 22118418
- [Background] Li WH, Chan SS, Wang KM, Lam TH. Helping cancer patients quit smoking by increasing their risk perception: a study protocol of a cluster randomized controlled trial. BMC Cancer. 2015 Jun 30;15:490. doi: 10.1186/s12885-015-1496-2. PMID 26122078
- [Background] Li WH, Wang MP, Lam TH, Cheung YT, Cheung DY, Suen YN, Ho KY, Tan KC, Chan SS. Brief intervention to promote smoking cessation and improve glycemic control in smokers with type 2 diabetes: a randomized controlled trial. Sci Rep. 2017 Apr 5;7:45902. doi: 10.1038/srep45902. PMID 28378764
- [Background] Abroms LC, Whittaker R, Free C, Mendel Van Alstyne J, Schindler-Ruwisch JM. Developing and Pretesting a Text Messaging Program for Health Behavior Change: Recommended Steps. JMIR Mhealth Uhealth. 2015 Dec 21;3(4):e107. doi: 10.2196/mhealth.4917. PMID 26690917
- [Background] Petty RE, Cacioppo JT. The elaboration likelihood model of persuasion. Adv Exp Soc Psychol. 1986;19:124-92.
- [Background] Stead LF, Perera R, Bullen C, Mant D, Lancaster T. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD000146. doi: 10.1002/14651858.CD000146.pub3. PMID 18253970
- [Background] Luo N, Liu G, Li M, Guan H, Jin X, Rand-Hendriksen K. Estimating an EQ-5D-5L Value Set for China. Value Health. 2017 Apr;20(4):662-669. doi: 10.1016/j.jval.2016.11.016. Epub 2017 Feb 9. PMID 28408009
- [Background] Lam TH, Abdullah AS, Chan SS, Hedley AJ; Hong Kong Council on Smoking and Health Smoking Cessation Health Centre (SCHC) Steering Group. Adherence to nicotine replacement therapy versus quitting smoking among Chinese smokers: a preliminary investigation. Psychopharmacology (Berl). 2005 Feb;177(4):400-8. doi: 10.1007/s00213-004-1971-y. Epub 2004 Jul 29. PMID 15289997
- [Background] Chan SS, Leung DY, Abdullah AS, Wong VT, Hedley AJ, Lam TH. A randomized controlled trial of a smoking reduction plus nicotine replacement therapy intervention for smokers not willing to quit smoking. Addiction. 2011 Jun;106(6):1155-63. doi: 10.1111/j.1360-0443.2011.03363.x. Epub 2011 Mar 7. PMID 21226883
- [Background] Lin PR, Zhao ZW, Cheng KK, Lam TH. The effect of physician's 30 s smoking cessation intervention for male medical outpatients: a pilot randomized controlled trial. J Public Health (Oxf). 2013 Sep;35(3):375-83. doi: 10.1093/pubmed/fdt018. Epub 2013 Mar 13. PMID 23487178
- [Background] Cromwell J, Bartosch WJ, Fiore MC, Hasselblad V, Baker T. Cost-effectiveness of the clinical practice recommendations in the AHCPR guideline for smoking cessation. Agency for Health Care Policy and Research. JAMA. 1997 Dec 3;278(21):1759-66. PMID 9388153
- [Background] Yudkin P, Hey K, Roberts S, Welch S, Murphy M, Walton R. Abstinence from smoking eight years after participation in randomised controlled trial of nicotine patch. BMJ. 2003 Jul 5;327(7405):28-9. doi: 10.1136/bmj.327.7405.28. No abstract available. PMID 12842953
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol. 2006;3(2):77-101.
- [Background] Michie S, Hyder N, Walia A, West R. Development of a taxonomy of behaviour change techniques used in individual behavioural support for smoking cessation. Addict Behav. 2011 Apr;36(4):315-9. doi: 10.1016/j.addbeh.2010.11.016. Epub 2010 Dec 15. PMID 21215528
- [Background] A clinical practice guideline for treating tobacco use and dependence: A US Public Health Service report. The Tobacco Use and Dependence Clinical Practice Guideline Panel, Staff, and Consortium Representatives. JAMA. 2000 Jun 28;283(24):3244-54. PMID 10866874
- [Background] Sabaté E. Adherence to long-term therapies: evidence for action. World Health Organization. 2003. Available from: http://apps.who.int/iris/bitstream/10665/42682/1/9241545992.pdf
- [Derived] Wu YS, Cheung YTD, Lee JJJ, Wong CKH, Ho SY, Li WHC, Yao Y, Lam TH, Wang MP. Effect of Adding Personalized Instant Messaging Apps to a Brief Smoking Cessation Model in Community Smokers in Hong Kong: Pragmatic Randomized Clinical Trial. J Med Internet Res. 2024 May 13;26:e44973. doi: 10.2196/44973. PMID 38739429